CLINICAL TRIAL: NCT02922192
Title: Incidence of Hospitalizations for Serious Infections in Patients Receiving Biologic Anti-Inflammatories for Rheumatologic, Psoriatic, and Gastrointestinal Conditions: A Descriptive Analysis
Status: Completed | Type: Observational
Sponsor: Biologics & Biosimilars Collective Intelligence Consortium (Other)
Collaborators: HealthCore, Inc. (Industry); Aetna, Inc. (Industry); University of Alabama; Rheumatologist and Healthcare Research (Unknown); AbbVie (Industry); Amgen (Industry); Boehringer Ingelheim (Industry); Kaiser Permanente (Other); Harvard Pilgrim Health Care (Other); Merck Sharp & Dohme LLC (Industry); Momenta Pharmaceuticals, Inc. (Industry); Pfizer (Industry); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: BBCIC-Anti-inflammatory
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis; Inflammatory Bowel Disease; Psoriasis; Psoriatic Arthritis; Ankylosing Spondylitis
Keywords: Anti-inflammatory; Biologics; Biologic and Biosimilars Collective Intelligence Consortium; BBCIC
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammatory Bowel Diseases; Psoriasis; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Rheumatoid arthritis (RA): With exposure to TNF-α antagonists, non-TNFs, DMARD non-biologics
  Interventions: Drug: TNF-α antagonists, non-TNFs, DMARD non-biologics
- Inflammatory bowel disease (IBD): With exposure to TNF-α antagonists, non-TNFs, DMARD non-biologics
  Interventions: Drug: TNF-α antagonists, non-TNFs, DMARD non-biologics
- Psoriatic conditions: Patients with a psoriasis, psoriatic arthritis, ankylosing spondylitis with exposure to TNF-α antagonists, non-TNFs, DMARD non-biologics
  Interventions: Drug: TNF-α antagonists, non-TNFs, DMARD non-biologics

INTERVENTIONS:
Drug: TNF-α antagonists, non-TNFs, DMARD non-biologics — Exposure to TNF- α antagonists, non-TNF- α antagonists, oral DMARD, or non-biologic agents.
  Other Names: 18 drug names in TNF, non-TNFs, DMARD non-biologics

SUMMARY:
Purpose:

With the existing biologic anti-inflammatory product patents expiring and the FDA approval of new biosimilar and innovator biologics, patients with rheumatologic (RA), psoriatic (PsO-PsA-AS), and gastrointestinal (GI) conditions will have additional therapeutic options. This observational study will describe the patient characteristics of new users of Tumor Necrosis Factor-α (TNF) antagonists, non-TNF- α antagonists, oral DMARD, and non-biologic agents. It will describe in the treatment cohorts outcomes of serious infections that require hospitalization. The BBCIC will use the findings from this descriptive analysis to design a comparative study evaluating the real-world effectiveness and safety of biosimilar and innovator anti-inflammatory biologics.

DETAILED DESCRIPTION:
Additional information:

To most effectively interpret results from this descriptive analysis it is important to consider that this protocol was not designed to support a hypothesis. This information is being provided to the public in the interest of transparency and for demonstrating the BBCIC's Distributed Research Network's (DRN) ability to define exposures, outcomes, covariates and confounders. When published, the report will caution that the protocol does not support any ability to compare safety or effectiveness but instead is to be used only to explore the feasibility of future, more detailed comparative analyses and to better understand the capabilities of the BBCIC project. Further, the report will caution that information from this protocol should not affect use of the medical products described in any way and the fact that the BBCIC is performing this descriptive analysis in no way suggests there is a safety or effectiveness issue with any of the products described.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with baseline period of 365 days with continuous medical and pharmacy coverage preceding the first prescription fill
* new and users of the following exposures

  * TNF -α antagonists (including adalimumab, certolizumab, etanercept [not included for IBD], golimumab, infliximab, and natalizumab [IBD only])
  * Non-TNF-alpha antagonist biologics in RA only (abatacept, rituximab, and tocilizumab)
  * Non-biologic medications (after any use of methotrexate in the previous year includes RA: hydroxychloroquine, leflunomide, or sulfasalazine; IBD: 6- mercaptopurine or azathioprine; PsO-PsA-AS: methotrexate, leflunomide, or sulfasalazine).

Exclusion Criteria:

* During baseline 365 days, any patient with

  * Active cancer or a history of non-melanoma cancer*
  * Any immunocompromising conditions (organ transplantation, HIV, and advanced kidney/liver disease)*
  * *if occur during the follow-up period, patients also will be censored.
* During baseline 183 days, any patient with hospitalization for any infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects are selected according to inclusion criteria from a source population within the Sentinel Common Data Mode v5.0.1 (SCDM). The SCDM includes over 100 million individuals with 358 million person-years of observation time who are covered by Aetna, Anthem, Group Health Cooperative, Harvard Pilgrim Health Care, and HealthPartners. The time period assessed will be 1/1/2006 - 9/30/2015.
Sampling Method: Non-Probability Sample
Enrollment: 90360 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hospitalization for serious infections | Anticipated completion January 2017
  Primary: Incidence of hospitalization for serious infections (i.e., infections of the respiratory tract, skin and soft tissue, genito-urinary tract, gastrointestinal tract, central nervous system, septicemia/sepsis).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Haynes, PharmD, MSCE, Principal Investigator — Anthem HealthCore, Inc.

IPD SHARING:
Plan to Share IPD: Yes
BBCIC Charter requires transparency and publication

REFERENCES:
- [Result] Mendelsohn AB, Nam YH, Marshall J, McDermott CL, Kochar B, Kappelman MD, Brown JS, Lockhart CM. Utilization patterns and characteristics of users of biologic anti-inflammatory agents in a large, US commercially insured population. Pharmacol Res Perspect. 2021 Feb;9(1):e00708. doi: 10.1002/prp2.708. PMID 33372729
- See also: The Biologics and Biosimilars Collective Intelligence Consortium (BBCIC) was established in 2015 to address anticipated needs for post-marketed evidence generation for novel biologics, their corresponding biosimilars and other related products. — http://www.bbcic.org